CLINICAL TRIAL: NCT06014151
Title: Study of the Motivations and Psychological Aspects of Gamete Donation Candidates Following the Change in the Law on Anonymity: a National Multicenter Study
Brief Title: Motivations and Psychological Aspects of Gamete Donation
Acronym: DONDON2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0272
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: GERM CELLS
Keywords: survey; gamete donation; motivations; psychological aspects; personality questionnaire; Neo-Pi-R; anonymat; sperm donation; oocyte donation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The candidate to gamete donation: All candidate to gamete donation at the CECOS centers in France
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — we will use a quantitative and a qualitative approach. For the first one, a psychosocial approach on a large number (500 women and 500 men) of candidates to donation. Of course, gender and parenthood will be considered in the analyses, as in the previous study. We will use two questionnaires for this study: 1) the one that was validated for the previous study, including socio-demographic data, donors' motivations and representations, 2) the second exploring personality, the NEO-PR inventory, which was also used for the previous study.

SUMMARY:
The objective of this project is to describe the motivations, the representation of donation and sterility, to evaluate the psychological aspects of the new male and female candidates to gamete donation and then to compare the results obtained from this population (post anonymity) with the previous population (anonymity).

DETAILED DESCRIPTION:
Context: The new bioethics law, August 2, 2021 introduced two major innovations: access to insemination with donor sperm without medical indication and access to the identity of the donor. This break in strict anonymity primarily concerns gamete donors. Countries where such a change has been made have often experienced a transitory decline in the number of donations and a change in the donor population. The centers feel that they are now receiving new donors. It will be important to monitor this evolution and to know the characteristics of the donors who will subsequently come in routinely, at a distance from the media episode generated by the discussions on the law.

In 2016-2018 we conducted a multicenter study on the motivations and psychological aspects of gamete donation. 20 centers were involved and the inclusion of 1021 gamete donation candidates allowed us to describe the motivations of these candidates, their representation of donation but also of infertility or family. We hypothesize that the new gamete donation candidates will be different in terms of their profile and their motivations. In this context we propose to conduct a study on the new population of gamete donation candidates but also to compare their characteristics with the previous population.

The objective of this project is to describe the motivations, the representation of donation and sterility, to evaluate the psychological aspects of the new male and female candidates to gamete donation and then to compare the results obtained from this population (post anonymity) with the previous population (anonymity).

The method. To do this, we will use a quantitative and a qualitative approach. For the first one, a psychosocial approach on a large number (500 women and 500 men) of candidates to donation. Of course, gender and parenthood will be considered in the analyses, as in the previous study. We will use two questionnaires for this study: 1) the one that was validated for the previous study, including socio-demographic data, donors' motivations and representations, 2) the second exploring personality, the NEO-PR inventory, which was also used for the previous study.

The second approach is qualitative through a clinical case study. It is a psychodynamic approach, which takes into consideration the female and male candidates to donation, with all their subjectivity, their personal and family history and their representations. 60 subjects, 30 donors versus 30 female donors, will be received for clinical interviews.

The data collected in this study will also be compared to the previous study, thus allowing to highlight the changes following the anonymity regime.

The expected results will allow a better understanding of the motivations of donors and to show the links of the latter with their parenthood status and gender and finally to evaluate the changes following the introduction of the possible access to the donor's identity. A better knowledge of these different points will be highly useful both for policy makers and information campaigns and for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All candidate to gamete donation at the CECOS centers in France

Exclusion Criteria:

* People who do not understand French or who cannot answer a paper questionnaire or an online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and men candidate to the gamete donation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of motivations and key personality traits through questionnaire data collection | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: NADJET NOURI, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France